CLINICAL TRIAL: NCT06206512
Title: A Crossover, Double-blinded, Two-period, Double Dummy Study to Evaluate the Effects of Extended Release Torsemide in Patients With Chronic Congestive Heart Failure and Symptoms of Overactive Bladder
Brief Title: Effect of Extended Release Torsemide in Patients With Congestive Heart Failure and Overactive Bladder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sarfez Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAR065-124
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Overactive Bladder; Incontinence
MeSH Terms: conditions — Heart Failure; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Crossover, double blinded, two-period, two-treatment, two-sequence, double dummy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Investigational product (Experimental): Extended release torsemide and immediate release torsemide placebo
  Interventions: Drug: Extended release torsemide; Drug: Immediate release torsemide placebo
- Control product (Active Comparator): Immediate release torsemide and extended release torsemide placebo
  Interventions: Drug: Immediate release torsemide; Drug: Extended release torsemide placebo

INTERVENTIONS:
Drug: Extended release torsemide — This is an extended-release formulation of torsemide
  Arms: Investigational product
Drug: Immediate release torsemide — This is the generic, immediate release formulation of torsemide
  Arms: Control product
Drug: Extended release torsemide placebo — Placebo of extended release torsemide
  Arms: Control product
Drug: Immediate release torsemide placebo — Placebo of immediate release torsemide
  Arms: Investigational product

SUMMARY:
This research study is being done to compare the effectiveness two drugs: an extended release torsemide (ERT) versus generic immediate release Torsemide (IRT) in reducing the worsening of symptoms of Overactive Bladder (OAB i.e., frequency, urgency, or urgency incontinence) in patients with chronic congestive heart failure (CHF).

This study will include CHF patients who experience worsening OAB) symptoms with use of a loop diuretic. The total duration of the study is about eight weeks with a total of nine visits.

There will be a screening visit that lasts one to two hours. The screening visit includes history and physical exams, blood draws, and urine analysis. If eligible for the study, participants will receive either generic torsemide or extended release torsemide for the first four weeks. Participants will do a virtual research visit on week one, two and three to submit a symptom diary and answer a questionnaire about urinary symptoms. At four weeks, history and physician exam will be done and blood will be collected. Participants will be assigned to receive either extended release torsemide (if they initially received generic torsemide) and generic torsemide (if they initially received extended release torsemide) for the next four weeks. Participants will attend virtual research visits on week five, six and seven to submit a symptom diary and answer a questionnaire about urinary symptoms. At the end of the study in week eight, they will have history and physical exams and blood draws.

Some risks from the study may include side effects of torsemide like acute kidney injury, fluid/electrolyte loss, hypersensitivity reactions and reversible hearing loss/tinnitus.

DETAILED DESCRIPTION:
This study has been designed to evaluate the efficacy of 24mg/48mg once daily dose of Investigational Product [Extended release torsemide of Sarfez Pharmaceuticals Inc.] to 20mg/40mg once daily dose of generic immediate release torsemide in reducing the symptoms of overactive bladder (OAB) in Chronic Heart Failure (CHF) patients.

Study Rationale Majority of chronic heart failure (CHF) patients are aged ≥50 and have symptoms of overactive bladder such as micturition frequency and urgency with or without urgency incontinence on stable dose of loop diuretics. Studies have shown that at normal physiological filling rate, intravesicular pressure does not rise until bladder capacity is reached. However, when the filling rate is higher than the normal physiological rate, the intravesicular pressure rises before bladder capacity is reached. Since loop diuretic increase filling rate, they are likely to raise intravesicular pressure much before it reaches capacity, and hence increase urgency. Therefore, there is a need for loop diuretic with a more gradual filling rate to alleviate loop diuretic induced exacerbation of symptoms OAB such as urgency and frequency. The proposed study follows upon successful clinical trial where in healthy volunteers, extended release torsemide of Sarfez Pharmaceutical Inc. decreased peak urine volume by >30% and induced gradual diuresis, indicating a gradual bladder filling. Therefore, this study is designed to determine if extended release torsemide of Sarfez Pharmaceutical Inc. can improve the bladder symptoms in heart failure patients as compared to a generic torsemide.

Patients who meet all inclusion and exclusion criteria, after obtaining written informed consent, will be screened using a four-question bladder condition assessment tool (score 0-5) and, only patients who score ≥4 score on each of the questions (total score ≥16) and meeting all other eligibility criteria will be enrolled in the study. The trial period will be divided into two periods as described above and shown in study flow schema (Figure 1). The total duration of the study would be 56 days excluding the day of enrolment in the study. Patients will visit the Clinical Research Unit/hospital at following schedules.

Visit 1: (Screening and Enrollment) start of study: After confirmation of eligibility and screening, patients will be randomized, HRQL tool and BS tool will be administered, (Baseline) and medications will be dispensed. Blood will be collected for NT-pro-BNP test and basic metabolic panel and body weight will also be measured. 6MWT will be performed. The other assessments will be done as mentioned in the study assessment schedule. Pregnancy test will be done to rule out pregnancy.

Period 1: All the enrolled patients who were on stable daily dose of furosemide will be randomized to either ERT or generic IRT. Patients who were on stable daily dose of furosemide 40 mg will be randomized to either ERT 24 mg or generic IRT 20 mg. Similarly, patients who were on stable daily dose of furosemide 80 mg will be randomized to either ERT 48 mg (two 24 mg tablets) or generic IRT 40 mg (two 20mg tablets). All pre-screening treatments will be recorded, and other concomitant medications will be continued (except non-steroidal anti-inflammatory agents but aspirin (<100 mg per day) will be permitted, cyclooxygenase-2 inhibitors such as Celecoxib, and allopurinol). On the same day HRQL tool and BS tool will be administered (Baseline assessments). Trained study coordinator will do a virtual visit on the last day of week 1, 2, and week 3 to provide and collect daily diary and to administer BS tool in week 2 and week 3. Upon diary collection, the study coordinator will check the diary for completion, and, if the diary is not properly completed, the study coordinator re-educates or re-instructs the patient with proper diary data filling procedures. Any retrospective modification or notation in the diary is strictly prohibited.

End of Period 1 and Cross Over: At the end of Week 4 (Day 28) patients will visit the site. After collecting daily diary from Period 1, the following assessment tools will be administered: HRQL tool, BS tool, and PGI-C questionnaires for frequency, urgency, urgency-incontinence, overall bladder problems, daily life and treatment satisfaction (anchors). Blood sample will be collected for basic metabolic panel and NT-proBNP and body weight will be measured. 6MWT will be performed along with physical examination and vital signs assessments.

On the same day medications will be switched and drug will be dispensed. Other assessments will be done as per the study assessment schedule.

Period 2: Trained study coordinator will do a virtual visit on the last day of week 5, week 6, and week 7 to provide daily diary and to collect the previous week's diary as well as to administer BS tool in week 6 and week 7. Upon diary collection, study coordinator will check the diary for completion, and, if the diary is not properly completed, the study coordinator will re-educate or re-instruct the patient with proper diary data filling procedures. Any retrospective modification or notation in the diary is strictly prohibited.

End of Study: At the end of Period 2 (Week 8, Day 56), following instruments will be administered along with the collection of weeks 8 diary: HRQL tool, BS tool, and PGI-C questionnaires for frequency, urgency, urgency-incontinence, overall bladder problems, daily life and treatment satisfaction (anchors). On the same day end of study assessment will be done as per the study assessment schedule and blood will be collected for basic metabolic panel and NT-pro-BNP. Also, body weight will be measured. 6MWT will be performed. End of study assessments will be performed as per study assessment schedule. Assessment Windows The deviations for the assessment times are acceptable based on logistical and operational considerations.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender of ≥50 years with clinical diagnosis of CHF.
* Patients with NYHA (New York Heart Association) functional class of II-IV
* Patients receiving stable dose of furosemide 40mg or 80mg daily for (>30 days).
* Patients with an estimated glomerular filtration rate (eGFR) of ≥30 ml/min/1.73 m2
* Patients with symptoms of overactive bladder

Exclusion Criteria:

* The patients with an estimated glomerular filtration rate (eGFR) below 30 ml/min/1.73 m2
* Requirement for a non-steroidal anti-inflammatory drug (NSAID), cyclooxygenase-2 (Cox-2) inhibitor (e.g., Celecoxib) or Allopurinol. If the patients are receiving these agents, they may be switched to acetaminophen, if agreed by the investigator and the dosing to be maintained throughout the study.
* Any known allergy to diuretics or sulphonamide-derived compounds
* Serum potassium concentration (K+) equal to or below 3.5 mEq/ L (mmol/L).
* History of myocardial infarction or stroke within the preceding 3 months duration
* Inability to comprehend or comply with the informed consent (including a physician's assessment of prior drug non-compliance).
* Urinalysis containing white blood cells indicative of urinary tract infection
* Patients with liver cirrhosis
* Any bladder catheterization, bladder, or prostrate surgery and/or, bladder, prostate, or pelvic radiotherapy within the last 3 months duration
* Patients who have participated in another clinical study in the past 3 months prior to commencement of this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Difference in average number of voiding, urgency, and urgency-incontinence episodes in the 2 groups | 56 days
  Assess the difference in average number of voiding, urgency, and urgency-incontinence episodes over 24 hours after dosing of Investigational product or Control product

SECONDARY OUTCOMES:
To assess the difference in average number of voiding, urgency, and urgency-incontinence episodes over 8 hours after dosing of IP or CP | 56 days
To assess the change in score from the baseline in bladder symptoms (BS Tool). | 56 days
To assess the change in scores from the baseline in overall health related quality of life and sub-scores (HRQL Tool). | 56 days
To assess the change in score from the baseline of Patient's Global Impression of Change (PGI-C) for frequency, urgency, urgency-incontinence, overall bladder problems, daily life, and treatment satisfaction | 56 days
To assess differences in the six-minute walk test (6MWT) scores between the treatment arms and from the baseline. | 56 days
To assess differences in the levels of NT-pro-BNP between the treatment arms and from the baseline | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Alvin Chandra, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Cardiometabolic Research Unit, Dallas, Texas, United States